CLINICAL TRIAL: NCT00548665
Title: Impact of Carotid Plaque Screening on Smoking Cessation and Control of Other Cardiovascular Risk Factors: A Randomized Controlled Trial.
Brief Title: Carotid Plaque Screening Trial in Smokers
Acronym: CAROSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Swiss National Science Foundation (Other); Swiss Heart Foundation (Other); Swiss Tobacco Prevention Funds (Unknown)
Responsible Party: Principal Investigator, Nicolas Rodondi, Prof. MD, MAS, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: SNSF 3200B0-116097
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Smoking
Keywords: Atherosclerosis; Smoking cessation; Diagnostic techniques, cardiovascular; Ultrasonography; Health behavior
MeSH Terms: conditions — Smoking; Atherosclerosis; Smoking Cessation; Health Behavior | interventions — Ultrasonography, Carotid Arteries; Crisis Intervention

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Carotid plaque screening and brief advice for smoking cessation: Smokers with at least one carotid plaque will receive pictures of their own plaques with a structured explanation on the general significance of plaques.
  Interventions: Device: Carotid ultrasound for plaque screening; Behavioral: Brief advice for smoking cessation
- 2 (Active Comparator): Brief advice for smoking cessation (without carotid ultrasound for plaque screening): to ensure equal contact conditions, smokers not undergoing ultrasound will receive a relevant explanation on the risks associated with tobacco smoking.
  Interventions: Behavioral: Brief advice for smoking cessation

INTERVENTIONS:
Device: Carotid ultrasound for plaque screening — Carotid ultrasound for plaque screening
  Other Names: B-mode ultrasound (Vingmed 5; General Electric Medical System, Wisconsin, USA), coupled with the M'ATH software (Metris, France).
  Arms: 1
Behavioral: Brief advice for smoking cessation — We will use the 5A's heuristic (Ask about smoking, Advise on cessation, Assess willingness to change, and for those willing to make quit attempt: Assist with attempt to quit, and Arrange for follow-up) and the gold standard for brief smoking cessation advice. At each visit, smokers will receive smoking cessation counseling and nicotine replacement therapy, similar to the experimental group.

SUMMARY:
The purpose of this study is to determine the impact of carotid plaque screening on smoking cessation and control of other cardiovascular risk factors.

DETAILED DESCRIPTION:
Tobacco smoking is highly prevalent in Switzerland (31% of adults), and 50% of smokers die from a tobacco-related disease, mainly cardiovascular disease (CVD). The smoking prevalence makes the evaluation of new strategies for smoking cessation a crucial priority.

The presence of plaques of atherosclerosis ("cholesterol" deposits in the artery wall), as measured by carotid ultrasound, increases the risk of future CVD. The use of plaque screening to motivate patients to improve smoking cessation has received little attention. In one study, screening for atherosclerotic plaques increased the self-reported rates of smoking cessation, but without biochemical validation of cessation and these smokers had only low nicotine dependence. Moreover, no trial has examined the impact of plaque screening on the control of other cardiovascular risk factors.

We now propose a randomized controlled trial of carotid plaque screening in 530 regular smokers aged 40-70 years, recruited from the community, to measure the impact of plaque screening on smoking cessation(main outcome) and control of other cardiovascular risk factors (secondary outcomes) after 1-year follow-up. Secondary outcomes are low-density lipoprotein cholesterol, hemoglobin A1C (if diabetes), high-sensitivity C-reactive protein and blood pressure. Smokers will all receive advice for smoking cessation and, then, will be randomly assigned to either the intervention group (with plaque screening) or the control group (without plaque screening). Smokers with one or more carotid plaque will receive pictures of their own plaques with a standardized explanation. To ensure equal contact conditions, smokers not undergoing ultrasound or without plaque will receive a standardized explanation on the risks of tobacco smoking.

This study is innovative because plaque screening is a promising and increasingly used strategy to motivate patients to stop smoking and improve control of cardiovascular risk factors, but its effectiveness has been poorly studied. Successful completion of this project will provide a strong scientific basis for using this strategy for smoking cessation and control of cardiovascular risk factors. If testing is not an effective tool, such testing might represent an important waste of expenditure, and healthcare expenditures should be used for other strategies. Given the scope of the global illness burden due to CVD, the simplicity of the proposed test (ultrasound of carotids) and the smoking prevalence in Switzerland, the evaluation of new strategies for smoking cessation in long-term smokers and the primary prevention of CVD is an important public health priority.

Beyond the randomized 1-year study, we have extended the follow-up to 3 years and added abdominal aneurysm screening by ultrasound to the intervention group to assess the association between cardiovascular risk factors and the development of small abdominal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Current daily smoker with more or equal to 10 cigarettes per day for at least 1 year
* Age between 40 and 70 years

Exclusion Criteria:

* Prevalent CVD at baseline, defined as a medical diagnosis or self-report of coronary heart disease, stroke or transient ischemic attack, peripheral arterial disease, carotid artery disease, congestive heart failure, or having a pacemaker.
* Unstable life-threatening or severe medical conditions (major arrhythmia, cancer,…)
* Current psychiatric disease
* Current substance abuse (cannabis, other drugs, alcohol abuse)
* Current use of pharmacological agent to quit smoking
* Current participation in another clinical trial
* Plan to move out of the French part of Switzerland in the following year
* Recent carotid ultrasound (< 1 year) to assess subclinical CVD
* Language barrier (not fluent with French)
* Potential difficulty to obtain good imaging of the carotid by ultrasound: past radiotherapy or major surgery of the neck

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence: one-week point prevalence abstinence, ascertained by self-report and confirmed by exhaled carbon monoxide (CO) and by the level of serum cotinine | 1 year, 3 years

SECONDARY OUTCOMES:
Continuous smoking abstinence from quit date and one-week point prevalence abstinence, ascertained by self-report and confirmed by exhaled carbon monoxide (CO) | 8 weeks, 26 weeks, 1 year, 3 years
Change in control of other cardiovascular risk factors: low-density lipoprotein cholesterol, hemoglobin A1C (if diabetes), high-sensitivity C-reactive protein (hs-CRP) and blood pressure. | 1 year, 3 years
Change in overall cardiovascular risk, as measured by the Framingham risk score | 1 year, 3 years
Change in drug adherence, as measured by adherence questionnaire | 1 year, 3 years
Change in quality of life, as measured by SF-36 | 1 year, 3 years
Change in physical activity, as measured by International Physical Activity Questionnaire questionnaire (IPAQ) | 1 year, 3 years
Increase in harms potentially associated with screening: stress and depression, as measured depression scores with the Beck Depression Inventory and the 4-item Perceived Stress Scale | 1 year, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, MD, MAS, Principal Investigator — University of Lausanne, Switzerland
Locations (1):
- University of Lausanne, Lausanne, Switzerland

REFERENCES:
- [Background] Rodondi N, Bovet P, Hayoz D, Cornuz J. The Impact of CAROtid plaque Screening on Smoking (CAROSS) cessation and control of other cardiovascular risk factors: Rationale and design of a randomized controlled trial. Contemp Clin Trials. 2008 Sep;29(5):767-73. doi: 10.1016/j.cct.2008.03.001. Epub 2008 Mar 18. PMID 18424239
- [Background] Rodondi N, Auer R, Devine PJ, O'Malley PG, Hayoz D, Cornuz J. The impact of carotid plaque screening on motivation for smoking cessation. Nicotine Tob Res. 2008 Mar;10(3):541-6. doi: 10.1080/14622200801902011. PMID 18324574
- [Result] Rodondi N, Collet TH, Nanchen D, Locatelli I, Depairon M, Aujesky D, Bovet P, Cornuz J. Impact of carotid plaque screening on smoking cessation and other cardiovascular risk factors: a randomized controlled trial. Arch Intern Med. 2012 Feb 27;172(4):344-52. doi: 10.1001/archinternmed.2011.1326. Epub 2012 Jan 23. PMID 22269590
- [Derived] Desgraz B, Collet TH, Rodondi N, Cornuz J, Clair C. Comparison of self-perceived cardiovascular disease risk among smokers with Framingham and PROCAM scores: a cross-sectional analysis of baseline data from a randomised controlled trial. BMJ Open. 2017 Jan 6;7(1):e012063. doi: 10.1136/bmjopen-2016-012063. PMID 28062468